CLINICAL TRIAL: NCT06337409
Title: A Single Dose, Randomized, Open-label, Two-way Crossover Bioequivalence Study of Generic Empagliflozin 25 mg Film-coated Tablets and Reference Product (JARDIANCE®) in Healthy Thai Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Empagliflozin 25 mg Film-coated Tablets in Healthy Thai Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: International Bio service (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BE24-004
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteer
Keywords: Empagliflozin 25 mg Film-coated Tablets
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin 25 mg film-coated tablets (Experimental): The test product, generic empagliflozin 25 mg film-coated tablets, will be formulated using the same active ingredient with the same strength as the reference product, JARDIANCE®. The test product to be used in this bioequivalence study is prepared in accordance with GMP regulations.
  Interventions: Drug: Generic empagliflozin 25 mg film-coated tablets
- Empagliflozin 25 mg film-coated tablets, JARDIANCE (Active Comparator): Empagliflozin 25 mg film-coated tablets, JARDIANCE®, has been registered with Food and Drug Administration, Thailand (TFDA).
  Interventions: Drug: Generic empagliflozin 25 mg film-coated tablets

INTERVENTIONS:
Drug: Generic empagliflozin 25 mg film-coated tablets — Empagliflozin 25 mg film-coated tablets
  Other Names: Empagliflozin

SUMMARY:
To determine and compare the rate and extent of absorption of a test formulation with that of a reference innovator formulation when given as equal labeled dose in healthy subjects under fasting conditions

DETAILED DESCRIPTION:
This study is conducted to investigate bioequivalence information which is required to ensure therapeutic equivalence of a test product and a reference product as well as to be considered as one aspect of product quality. Bioequivalence is defined as the absence of a significant difference in the rate and extent to which the active ingredient or active moiety in pharmaceutical equivalents or pharmaceutical alternatives becomes available at the site of drug action when administered at the same molar dose under similar conditions in an appropriately designed study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Thai male or female subjects between the ages of 18 to 55 years
* Body mass index between 18.5 to 30.0 kg/m2.
* Normal laboratory values, including vital signs and physical examination, for all parameters in clinical laboratory tests at screening. Any abnormalities from the normal or reference range will be carefully considered clinically relevant by the physician as individual cases, documented in study files prior to enrolling the subject in this study
* Non-pregnant woman (negative pregnancy test) and not currently breast feeding
* Female subjects abstain from either hormonal methods of contraception (including oral or transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) or hormone replacement therapy for at least 28 days prior to check-in in Period 1. Injectable contraceptives e.g. Depo-Provera® will be discontinued at least 6 months prior to check-in in Period 1. Subjects agree to use acceptable non-hormonal contraceptive methods such as condom, diaphragm, foams, jellies, or abstinence for at least 14 days prior to check-in in Period 1 until 7 days after the end of study in Period 2. Female subjects of non-childbearing potential must meet at least one of the following criteria prior to check-in in Period 1:
* Postmenopausal for at least 1 year or
* Surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) at least 6 months
* Male subjects who are willing or able to use effective contraceptive e.g. condom or abstinence after check-in in Period 1 until 7 days after the end of study in Period 2.
* Have voluntarily given written informed consent (signed and dated) by the subject prior to participating in this study

Exclusion Criteria:

* History of allergic reaction or hypersensitivity to empagliflozin or to any of the excipients.
* History or evidence of clinically significant renal, hepatic, gastrointestinal, hematological (e.g. anemia), endocrine (e.g. hyper/hypothyroidism, diabetes mellitus), pulmonary or respiratory (e.g. asthma), cardiovascular (e.g. hyper/hypotension), psychiatric (e.g. depression), neurologic (e.g. seizures), allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or any significant ongoing chronic medical illness.
* Have high risk for coronavirus infection based on risk assessment questionnaire or diagnosed as confirmed case of COVID-19.
* History about administration of COVID-19 vaccine within 30 days prior to check-in in each Period.
* Investigation with blood sample shows fasting blood glucose level less than 70 mg/dl or more than 99 mg/dl at screening
* History or evidence of type 1 diabetes mellitus or diabetic ketoacidosis.
* History or evidence of heart failure.
* History or evidence of volume depletion or hypotension.
* History or evidence of genital mycotic infections, urinary tract infections within 14 days prior to check-in in each period.
* History or evidence of necrotizing fasciitis of the perineum (fournier's gangrene).
* History or evidence of galactose intolerance, the Lapp lactase deficiency or glucosegalactose malabsorption
* History of problems with swallowing tablet or capsule.
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Any condition possibly affecting drug absorption e.g. gastrectomy, enterectomy, gastritis or duodenal or gastric ulceration other than appendectomy.
* History of diarrhea or vomiting within 24 hours prior to check-in in each period
* History or evidence of drug addict or investigation with urine sample shows a positive test for drug of abuse (morphine, marijuana or methamphetamine).
* Investigation with blood sample shows positive test for HBsAg
* Abnormal liver function, ≥1.5 times of upper normal limit of reference range for ALT, AST or bilirubin levels at screening laboratory test
* Have eGFR (CKD-EPI) < 45 mL/min/1.73 m2 based on serum creatinine results, at the screening laboratory test or during enrollment.
* History or evidence of habitual use of tobacco or nicotine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study
* History or evidence of alcoholism or harmful use of alcohol (less than 2 years) i.e., alcohol consumption of more than 14 standard drinks per week for men and 7 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 mL of 40% distilled spirits, such as rum, whisky, brandy, etc.).
* History or evidence of alcohol consumption or alcohol-containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study or alcohol breath test shows positive result. In case of alcohol breath test result represents the alcohol concentration range of 1-10 mg% BAC and the physician carefully considers that the value came from other reasons, not from the alcohol drinking behavior of subjects, the test will be repeated two times separately, not more than 10 minutes. The result of the last time should be used for subject's eligibility which must be 0 mg%BAC.
* History or evidence of habitual consume of tea, coffee, xanthine or caffeine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study.
* Consume or drink juice of grapefruit or orange or pomelo or its supplement/containing products and cannot abstain for at least 7 days prior to check-in in Period 1 and continued for entire duration of the study.
* Use of prescription or nonprescription drugs (e.g. paracetamol, lithium, digoxin, warfarin, verapamil, ramipril, simvastatin, gemfibrozil, rifampicin, probenecid, insulins, insulin secretagogues, other antidiabetics and diuretic drugs), herbal medications or supplements (e.g. St. John's wort), vitamins or mineral (e.g. iron) or dietary supplements within 14 days prior to check-in in Period 1 and continued for entire duration of the study.
* Participated in other clinical trials within 90 days prior to check-in in Period 1 (except for the subjects who drop out or withdrawn from the previous study prior to Period 1 dosing) or still participates in the clinical trial or participates in other clinical trials during enrollment in this study.
* Blood donation or blood loss ≥ 1 unit (1 unit is equal to 350-450 mL of blood) within 90 days prior to check-in in Period 1 or during enrollment.
* Subjects with poor venous access or intolerant to venipuncture
* Unwilling or unable to comply with schedule visit, treatment plan and other study procedures until end of study.
* Inability to communicate well (i.e. language problem, poor mental development, psychiatric illness or poor cerebral function) that may impair the ability to provide written informed consent or cooperate with clinical team.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-07-05 (Estimated); Study Completion 2024-07-13 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax period | Through 72 Hours Post Dose
  Bioequivalence based on Cmax period

SECONDARY OUTCOMES:
Bioequivalence based on AUC parameters | Through 72 Hours Post Dose
  Bioequivalence based on AUC parameters

CONTACTS AND LOCATIONS:
Overall Officials: Uthai Suvanakoot, Ph. D, Principal Investigator — International Bio service

IPD SHARING:
Plan to Share IPD: No
Confidential